CLINICAL TRIAL: NCT02028182
Title: Clinical Evaluation of Hydroxyisohexyl 3-cyclohexene Carboxaldehyde (Lyral®) Dose Response Study
Brief Title: Clinical Evaluation of Lyral® Dose Response Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allerderm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12 1PL 201
Record Dates: First submitted 2014-01-02; First posted 2014-01-07 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2014-01

CONDITIONS: Contact Dermatitis
Keywords: Patch Test; Allergy Testing; Contact dermatitis; Lyral allergen; Fragrance Mix allergen
MeSH Terms: conditions — Dermatitis, Contact | interventions — hydroxyisohexyl 3-cyclohexene carboxaldehyde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Positive reactions, Concordance with reference allergen (Experimental): Subjects were patch tested with an experimental allergen panel containing ascending doses of Lyral (0.10 mg/cm2, 0.20 mg/cm2 and 0.40 mg/cm2) and a negative control. A second panel containing 20 mg of 5% Lyral in petrolatum was applied for evaluation of concordance. The panels were worn for approximately 48 hours. Skin reactions were assessed at 3, 4 and 21 days following application.
  Interventions: Biological: Lyral®

INTERVENTIONS:
Biological: Lyral® — Alergen panel containing ascending doses of Lyral (0.10 mg/cm^2, 0.20 mg/cm^2 and 0.40 mg/cm^2) and negative control
  Other Names: Lyral Allergen Panel (experimental)

SUMMARY:
The purpose of this study is to determine optimal allergen dose as the lowest concentration eliciting positive reactions in 70-90% of subjects. Frequency of positive, negative, doubtful and irritant reactions, and concordance with a corresponding reference allergens will be captured.

DETAILED DESCRIPTION:
This is a single-center, randomized study to compare the diagnostic performance and safety of ascending doses (0.10 mg/cm², 0.20 mg/cm² and 0.40 mg/cm²) of hydroxyisohexyl 3-cyclohexene carboxaldehyde (Lyral®) in 20 adult subjects with a past positive patch test to Lyral® or Fragrance Mix 2.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age and older.
2. Clinical history of contact dermatitis and positive patch test (current or previous) to either Lyral® or Fragrance Mix 2; otherwise in good general health.
3. Unable to become pregnant or willing to use an acceptable method of contraception to prevent pregnancy if female of childbearing potential; Inability to become pregnant would include all male subjects and female subjects who are postmenopausal for at least 1 year, or surgically sterile- have had a hysterectomy, bilateral ovariectomy, uterine ablation or bilateral tubal ligation.

   Acceptable methods of contraception include: 1) systemic birth control (the same type of birth control for at least 3 months prior to entering the study and continuation of this type of birth control throughout the study); 2) double barrier methods (condom with spermicide or diaphragm with spermicide); 3) intra uterine device; 4) vasectomized partner; or 5) abstinence from sexual intercourse.
4. Have read and signed the consent form and are able to fulfill the study requirements and make all required visits.

Exclusion Criteria:

1. Lactation or pregnancy, determined by urine pregnancy test (UPT) for females of childbearing potential. UPT must be conducted prior to patch placement.
2. Treatment with topical corticosteroids on or near the test area during the previous 7 days.
3. Treatment with systemic corticosteroids or immunosuppressives during the previous 7 days. (Inhaled treatments are permitted.)
4. Treatment with ultraviolet (UV) light, including tanning, during the previous 3 weeks.
5. Acute dermatitis outbreak or dermatitis on or near the test area on the back.
6. Participation in another clinical study involving an investigational drug, treatment or device currently or within the previous 3 weeks.
7. Unable to comply with activity restrictions (e.g., protecting test panels from excess moisture due to showering or vigorous activity).
8. Unable or unwilling to comply with multiple return visits.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evy Paulsen, Md, PhD, Principal Investigator — Department of Dermatology and Allergy Centre Odense University Hospital
Locations (1):
- University of Southern Denmark Institute of Clinical Research, Odense, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Positive Reactions, Concordance With Reference Allergen: Subjects were patch tested with an experimental allergen panel containing ascending doses of Lyral (0.10 mg/cm^2, 0.20 mg/cm^2 and 0.40 mg/cm^2) Lyral® and a negative control. A second panel containing 20 mg of the marketed Lyral allergen, 5%, in petrolatum was applied for evaluation of concordance. The panels were worn for approximately 48 hours. Skin reactions were assessed at 3, 4 and 21 days following application.
  Lyral®: T.R.U.E. Test allergen panel containing ascending doses of Lyral (0.10 mg/cm^2, 0.20 mg/cm^2 and 0.40 mg/cm^2) and negative control
Period: Overall Study
Arm/Group | Positive Reactions, Concordance With Reference Allergen
Started | 22
Completed | 20
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- Positive Reactions, Concordance With Reference Allergen: Subjects were patch tested with an experimental allergen panel containing ascending doses of Lyral (0.10 mg/cm2, 0.20 mg/cm2 and 0.40 mg/cm2) and a negative control. A second panel containing 20 mg of 5%, in petrolatum was applied for evaluation of concordance. The panels were worn for approximately 48 hours. Skin reactions were assessed at 3, 4 and 21 days following application.
  Allergen panel containing ascending doses of Lyral (0.10 mg/cm2, 0.20 mg/cm2 and 0.40 mg/cm2) and negative control
Arm/Group | Positive Reactions, Concordance With Reference Allergen
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 5
Region of Enrollment [Number; unit: participants]
  Denmark | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Patch Test Responses
Description: Subjects were patch tested with one experimental T.R.U.E. Test allergen panel containing 0.40 mg/cm^2, 0.20 mg/cm^2, and 0.10 mg/cm^2 of Lyral® and a negative control and a second panel containing the marketed reference allergen (20 mg of Lyral® 5%, in petrolatum). The panels were worn for approximately 48 hours. Skin reactions were assessed at 3, 4 and 21 days following application. Negative responses are graded no response, doubtful response (faint erythema, no infiltration), or irritant response (patchy erythema, no infiltration). Positive responses are graded 1+ (erythema, infiltration, discrete papules), 2+ (erythema infiltration, papules, discrete vesicles), or 3+ (coalescing vesicles, bullous reaction)
Time Frame: Patch test sites were evaluated at day 3 or 4, day 7 and day 21 following application. Results were assessed by the Investigator following the day 21 visit.
Measure: Number; unit: participants
Arm/Group | Positive Reactions, Concordance With Reference Allergen
Number analyzed (Participants) | 20
participants
  0.40 mg/cm^2 Lyral Positive Responses | 14
  0.20 mg/cm^2 Lyral Positive Responses | 12
  0.10 mg/cm^2 Lyral Positive Responses | 11
  Negative Control Positive Responses | 0
  0.40 mg/cm^2 Lyral Negative Responses | 6
  0.20 mg/cm^2 Lyral Negative Responses | 8
  0.10 mg/cm^2 Lyral Negative Responses | 9
  Negative Control Negative Responses | 20
Statistical Analysis 1: Comparison: Positive Reactions, Concordance With Reference Allergen; Test type: Other; Kappa statistic-Concordance 0.4 mg/cm2 = 75.0, 95% CI 2-sided [60.4 to 94.0]
Statistical Analysis 2: Comparison: Positive Reactions, Concordance With Reference Allergen; Test type: Other; Kappa statistic: Concordance 0.20 mg/cm2 = 65.0, 95% CI 2-sided [55.6 to 90.4]
Statistical Analysis 3: Comparison: Positive Reactions, Concordance With Reference Allergen; Test type: Other; Kappa statistic: Concordance0.10 mg/cm2 = 60.0, 95% CI 2-sided [53.3 to 88.4]

2. Secondary Outcome: Number of Subjects With Tape Irritation, Itching and Burning
Description: Tape irritation is graded on a 4 point scale: None (no tape irritation), Weak (faint to definite pink), Moderate (moderate erythema, definite redness) and Strong (severe erythema, very intense redness). Percentage of response will include weak, moderate and strong reactions.
  Itching and Burning are graded on a 4 point scale: None (no discomfort), Weak (minimal discomfort), Moderate (definite discomfort) and Strong (significantly bothersome, possible interference with sleep or daily activity). Percentage of response will include weak, moderate and strong responses.
Time Frame: Day 2: 48 hours after application
Measure: Number; unit: participants
Arm/Group | Positive Reactions, Concordance With Reference Allergen
Number analyzed (Participants) | 22
participants
  Tape Irritation: None | 14
  Tape Irritation: Weak | 8
  Tape Irritation: Moderate | 0
  Tape Irritation: Strong | 0
  Itching: None | 7
  Itching: Weak | 10
  Itching: Moderate | 4
  Itching: Strong | 1
  Burning: None | 17
  Burning: Weak | 3
  Burning: Moderate | 2
  Burning: Strong | 0

3. Secondary Outcome: Number of Subjects Who Exhibit Late or Persistent Reactions
Description: Late reactions initially occur at 7-21 days after application of the panels Persistent reactions appear at Day 2-4 and persist through Day 7-21
Time Frame: Days 2-21
Measure: Count of Participants; unit: Participants
Arm/Group | Positive Reactions, Concordance With Reference Allergen
Number analyzed (Participants) | 20
Participants
  0.40 mg/cm^2 Late Reactions | 1
  0.20 mg/cm^2 Late Reactions | 1
  0.10 mg/cm^2 Late Reactions | 2
  0.40 mg/cm^2 Persistent Reactions | 13
  0.20 mg/cm^2 Persistent Reactions | 10
  0.10 mg/cm^2 Persistent Reactions | 7

ADVERSE EVENTS:
Time Frame: Days 2-21
Groups:
- Positive Reactions, Concordance With Reference Allergen: Subjects were patch tested with an experimental allergen panel containing all doses of Lyral (0.10 mg/cm^2, 0.20 mg/cm^2 and 0.40 mg/cm^2) Lyral® and a negative control. A second panel containing 20 mg of the marketed Lyral allergen, 5%, in petrolatum was applied for evaluation of concordance. It is not possible to discern specific dose relative to adverse events.
Arm/Group | Positive Reactions, Concordance With Reference Allergen
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 3/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Positive Reactions, Concordance With Reference Allergen (N=22)
Conjunctivitus (Eye disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No